CLINICAL TRIAL: NCT05544227
Title: Immunotherapy Regimen Given After Targeted Local Cryolysis (TLC) for Patients With Advanced/Metastatic Castration-resistant Prostate Cancer (mCRPC) OR Those With Metastatic Prostate Cancer Who Refused Hormone Therapy and Chemotherapy.
Brief Title: Phase 1 Trial of SYNC-T - Immunotherapy for Advanced/Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Williams Cancer Foundation (Other)
Collaborators: Syncromune, Inc. (Industry)
Responsible Party: Principal Investigator, Carlos Vargas, MD, Principal Investigator, Williams Cancer Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phase 1 SV-102
Record Dates: First submitted 2022-08-16; First posted 2022-09-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SV-102 Treatment Arm (Experimental): SV-102 Treatment Arm
  Interventions: Drug: SV-102

INTERVENTIONS:
Drug: SV-102 — SV-102 is intended to overcome the complex and multifactorial nature of the mechanisms mediating tumor immune evasion, by the use of a combination of therapeutic agents that elicit multiple immunopharmacologic effects.

SUMMARY:
SV-102 is intended to overcome the complex and multifactorial nature of the mechanisms mediating tumor immune evasion, by the use of a combination of therapeutic agents that elicit multiple immuno-pharmacologic effects.

DETAILED DESCRIPTION:
SV-102 is intended for immunotherapeutic treatment of solid tumors in certain metastatic cancer indications. SYNC-T™ technology encompasses methods and compositions that mediate multiple pharmacologic effects aimed at mounting a synchronized and multi-faceted antitumor immune response. The first component of SYNC-T™ is aimed at eliciting in situ immunization by triggering the lysis and immunogenic cell death of tumor cells, followed by the release of tumor-specific or tumor-associated antigens (TSA/TAAs) and danger associated molecular patterns (DAMPs) into the tumor microenvironment. The main approach that will be used by SYNC-T™ will rely on partial and targeted local cryolysis of tumor cells mediated by a cryolysis device. The second component of SYNC-T™ technology is the intratumoral infusion of a low-dose multi-component drug product.

ELIGIBILITY:
Inclusion Criteria:

1. Male >18 years old at the time of signed informed consent
2. Provide written informed consent
3. Subjects with advanced and/or metastatic histologically or cytologically confirmed castrate-resistant prostate cancer
4. After failure after the receipt of previous treatment with one or more approved second-generation androgen-receptor-pathway inhibitors and with or without a prior course of taxanes therapy or those with metastatic prostate cancer who have refused hormone therapy and chemotherapy, or have not responded or progressed after standard therapies or for whom no further standard therapy exists or standard therapy is not available
5. Patients who may or may not have had prior therapy with Lutetium Lu-177-PSMA-I&T
6. Resolution of all acute toxic effects (excluding alopecia) of any prior anti-cancer therapy to National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) v5 grade ≤ 1.
7. Measurable disease by RECIST.
8. Meet all eligibility criteria
9. Able to undergo general anesthesia or conscious sedation
10. Has undergone a cardiac work-up and received cardiac clearance two months before first treatment
11. Has halted use of any anticoagulants or other blood thinners (including but not limited to heparin or warfarin) within five (5) days of each treatment.
12. Eastern Cooperative Oncology Group (ECOG) performance status of < 3 (0, 1, or 2)
13. All subjects with female partners of childbearing potential must use effective contraception throughout study treatment and for 120-150 days (4-5 months) after the last dose of study intervention
14. Has at least one lesion within the prostate accessible transperineally using transrectal ultrasound (TRUS) that is demonstrable on PET/CT, CT, Ultrasound, or MRI and is accessible for infusion on TRUS or, if a radical prostatectomy has been performed, has a metastatic lesion or lymph node lesion that is demonstrable on PET/CT, CT, or MRI and accessible by a percutaneous needle to permit treatment.
15. Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must be on stable doses for at least 42 days prior to the cryolysis
16. Adequate bone marrow, renal, and hepatic function, defined as follows:

    a. Bone marrow function without transfusion 30 days before first dosing: i. Absolute neutrophil count ≥ 1.5 x 109/L; Lymphocyte count of ≥ 1.0 x 109/L; Platelet count ≥ 100 x 109/L; ii. Hemoglobin ≥ 9.0 g/dL b. Renal function" i. Estimated glomerular filtration rate ≥30 mL/min/1.73 m2 or creatinine clearance calculated by Cockcroft-Gault equation ≥30 mL/ c. Hepatic function i. Alanine aminotransferase ≤ 3x upper limit of normal (ULN) ii. Aspartate aminotransferase ≤ 3x ULN iii. Total bilirubin ≤ ULN or total bilirubin ≤ 1.5x ULN with direct bilirubin ≤ ULN of the laboratory in subjects with documented Gilbert's Syndrome iv. Patients with liver metastases ≤5x ULN
17. All clinically relevant toxicities related to prior anticancer therapy must have recovered to Grade ≤1 or baseline (except alopecia or ototoxicity

Exclusion Criteria:

1. Has a known other primary malignancy other than prostate cancer that is progressing or has required active treatment in the last 3 years, excluding basal and squamous cell carcinoma, papillary thyroid cancer, and ductal carcinoma in situ of the breast
2. Has an obstructed urinary system before or after stenting
3. Has undergone major surgery, including local prostate intervention (excluding prostate biopsy), within 28 days prior to the first dose of study drug and has not recovered adequately from the toxicities and/or complications
4. Has an active infection (including tuberculosis) requiring systemic therapy
5. Has a history of non-infectious pneumonitis that required steroids
6. Has received a live vaccine within 30 days prior to the enrollment Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 28 days prior to the first treatment
7. Significant cardiac or other medical illness such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia (e.g. New York Heart Association Class 4), or history of previous heart failure
8. Malignant pleural effusions or ascites that require immediate intervention
9. Prior history of autoimmune disease except hypothyroidism, uncontrolled or unmanaged diabetes, cardiac arrhythmia (unstable or untreated), hypersensitivity, or other illness or disease that in the opinion of the Principal Investigator, with consultation with Syncromune's Chief Medical Officer, makes the subject a poor candidate.
10. Any primary or acquired immunodeficiency
11. Active COVID infection or tests positive for COVID day before or day of planned treatment
12. Known or suspected hepatitis B if active infection (subjects with chronic hepatitis B infection must have an undetectable Hepatitis B virus (HBV) viral load on suppressive therapy, if indicated; positive surface antibody alone is not an exclusion)
13. Known or suspected hepatitis C infection which has not been treated and cured unless currently on treatment with an undetectable viral load
14. Any condition(s) that, in the opinion of the Investigator, would increase the risk for toxicities from study drug, interfere with subject compliance or conduct of this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Baseline through 30 days after end-of-treatment
  Summary of treatment-emergent AEs, including NCI CTCAE v5.0 severity grade and relationship to either the device or study drugs.
Number of participants with deaths | Baseline through 30 days after end-of-treatment
  Summary of deaths leading to study discontinuation
Number of participants with treatment-emergent SAEs and AEs | Baseline through 30 days after end-of-treatment
  Summary of treatment-emergent SAEs, and AEs leading to study discontinuation
Assessment of laboratory values. | Baseline through 30 days after end-of-treatment
  Summary of laboratory values over time and shifts in laboratory measurements by NCI CTCAE v5.0 grade.

SECONDARY OUTCOMES:
Number of patients in the Intent-to-Treat Population with complete response to SV-102. | Baseline through 12 weeks after end-of-treatment
  Summary of objective response rate (ORR), presented as the percentage of patients with a complete response as assessed by the Investigator using PCWG3.
Number of patients in the Intent-to-Treat Population with complete response to SV-102. | Baseline through 12 weeks after end-of-treatment
  Summary of objective response rate (ORR), presented as the percentage of patients with a complete response as assessed by the Investigator using RECIST 1.1.
Number of patients in the Intent-to-Treat Population with complete response to SV-102. | Baseline through 12 weeks after end-of-treatment
  Summary of objective response rate (ORR), presented as the percentage of patients with a complete response as assessed by the Investigator using iRECIST.
Number of patients in the Intent-to-Treat Population with partial response to SV-102. | Baseline through 12 weeks after end-of-treatment
  Summary of objective response rate (ORR), presented as the percentage of patients with a partial response as assessed by the Investigator using PCWG3.
Number of patients in the Intent-to-Treat Population with partial response to SV-102. | Baseline through 12 weeks after end-of-treatment
  Summary of objective response rate (ORR), presented as the percentage of patients with a partial response as assessed by the Investigator using RECIST 1.1.
Number of patients in the Intent-to-Treat Population with partial response to SV-102. | Baseline through 12 weeks after end-of-treatment
  Summary of objective response rate (ORR), presented as the percentage of patients with a partial response as assessed by the Investigator using iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vargas, MD, Principal Investigator — Williams Cancer Institute
Locations (1):
- Hospital Diomed, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No